CLINICAL TRIAL: NCT02034305
Title: Pilot Study of Cough Peak Flow And Airway Clearance in Pediatric Patients With Neuromuscular Disease
Brief Title: Peak Cough Flow and Cough Clearance in Patients With Muscular Dystrophy
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Respirtech, Inc. (Industry)
Responsible Party: Principal Investigator, Daniel J. Weiner, Associate Professor of Pediatrics, University of Pittsburgh
Other Study IDs: PRO11100704
Record Dates: First submitted 2014-01-09; First posted 2014-01-13 (Estimated); Last update posted 2024-02-05 (Actual); Status verified 2021-01

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Airway Clearance; Duchenne Muscular Dystrophy; Peak Cough Flow
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study is to determine whether physiologic measures (peak cough flow, measures of respiratory muscle strength including MIP, MEP ,SNIP, and spirometry) can predict spontaneous cough clearance (as measured by a nuclear medicine study) in children with neuromuscular disease. It will also determine whether airway clearance is augmented by high frequency chest wall oscillation.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-21; able to cooperate with study procedures
* Duchenne Muscular Dystrophy OR Becker Muscular Dystrophy

Exclusion Criteria:

* Need for mechanical ventilation during the day
* Recent (within 2 weeks) lower respiratory tract infection

Ages: 6 Years to 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Boys 6-21 years of age with Duchenne Muscular Dystrophy
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2014-01; Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Spontaneous cough clearance | Assessed at multiple time points over 30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Weiner DJ, Abdel-Hamid H, Corcoran TE. Pilot study of nuclear scintigraphy to assess cough clearance in DMD. Pediatr Pulmonol. 2022 Jul;57(7):1776-1778. doi: 10.1002/ppul.25894. Epub 2022 May 5. No abstract available. PMID 35293696